CLINICAL TRIAL: NCT06200857
Title: Impact of Socioeconomic and Territorial Inequalities on Surgical Management of Sigmoid Diverticulitis: French National Multicenter Retrospective Study
Brief Title: Impact of Socioeconomic and Territorial Inequalities on Surgical Management of Sigmoid Diverticulitis
Acronym: EDIVERTICULITE
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 20-510
Record Dates: First submitted 2023-12-20; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Sigmoid Diverticulosis; Colorectal Surgery
Keywords: sigmoid diverticulitis _ surgery _ socio-economic inequalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- association francaise de chirurgie AFC working group: cohort description included all patients aged over 18, undergoing emergency or elective surgery for sigmoid diverticulitis between 2010 and 2019 and with a follow-up of at least 3 months to determine morbi-mortality on the 90th postoperative day.
  minor patient, those with a final colorectal cancer and those operated on for right colonic diverticulitis were excluded
  with a follow-up of at least 3 months to determine morbi-mortality on the 90th postoperative day.
  Non-inclusion criteria for research subjects :
  * Minor patient
  * Surgical finding of colorectal cancer The patient operated on for diverticulitis of the right colon

SUMMARY:
Sigmoid diverticulitis (SD) is a common pathology characterized by inflammation/infection of a diverticulum in the sigmoid colon. Surgical treatment of DS is indicated urgently, either because of a serious complication or because of therapeutic failure. Prophylactic surgical treatment of "cold" DS is indicated in symptomatic forms (smoldering diverticulitis, frequent recurrences impacting quality of life, symptomatic fistula, and stenosis). It is also indicated for asymptomatic forms in selected patients, to avoid recurrence and/or the occurrence of a DS complication. In France, some 12,000 prophylactic colectomies for DS are performed every year. The mortality rate for this operation during the hospital stay (which does not account for 30-day mortality) is 7 per thousand in France. Morbidity is fairly high, at around 25%, with almost 10% of severe complications. At a distance, the definitive stoma rate is around 6% of patients, and recurrences have been described in up to 10% of cases. Numerous clinical determinants linked to the patient and the pathology have been identified as potential risk factors for morbidity and mortality (advanced age, undernutrition, emergency surgery, neurological history, minimally invasive approach, etc.). Among non-clinical determinants, socio-economic and territorial deprivation is thought to have an impact on postoperative morbidity and mortality for a very large number of pathologies, including cardiovascular disease, cancer, and obesity. Thus, patients from the most disadvantaged backgrounds would have a significantly higher risk of postoperative mortality and morbidity. To our knowledge, however, few data are available on the possible impact of socio-economic deprivation and geographical isolation on the operative outcome of colorectal surgery. This French multicenter study aims to assess the impact of socio-economic and territorial inequalities on the surgical management of sigmoid diverticulitis; with the primary objective being the prevalence of postoperative complications and the secondary objectives being the prevalence of recourse to emergency surgery, minimally invasive surgery, definitive stoma and post-operative recurrence.

DETAILED DESCRIPTION:
Surgical treatment of sigmoid diverticulitis (SD) is indicated as an emergency measure, either immediately in the event of a serious complication or secondarily in the event of therapeutic failure.

New French recommendations for prophylactic surgery have been published since 2017. Systematic elective sigmoidectomy after acute diverticulitis attack is not recommended if the patient is asymptomatic, not immunocompromised or chronically renal-impaired, and if attack does not impact the quality of life (Grade B). Elective sigmoidectomy is recommended in the following situations: (i) after complicated acute diverticulitis, particularly in the case of abscesses; (ii) in immunocompromised patients or those with chronic renal insufficiency, taking into account the following operative risk factors (age over 75 and comorbidities, particularly heart disease and COPD) (Grade C). In asymptomatic patients, age under 50 does not in itself constitute an indication for surgery (Grade B). It is recommended to propose elective sigmoidectomy in cases of persistent symptoms after a relapse (including smoldering diverticulitis) or frequent recurrences affecting quality of life. The number of relapses is not an indication in itself (Grade C). Elective sigmoidectomy is recommended in cases of fistula, depending on the terrain and type of symptoms. Elective sigmoidectomy is recommended in cases of symptomatic stenosis (grade C).

These updated recommendations aimed to improve the management of patients with SD through more appropriate surgical procedures and to harmonize professional practices. They are all the more relevant in that it is estimated that nearly 12,000 prophylactic colectomies for SD are performed each year in France.

Mortality after prophylactic colectomy for SD is documented by two national databases. In the 1st database, representing 20% of US national data from 2003 to 2009, 74,879 patients underwent colectomy either for SD (50.52%), colon cancer (43.48%), or inflammatory disease (6.00%). In-hospital mortality after prophylactic colectomy for SD was 0.4% (15). After adjustment for age, gender, ethnicity, period of admission, and Charlson comorbidity score, compared with colon cancer, colectomy for SD was associated with an excess risk of mortality (adjusted OR (AOR)= 1.9 IC95%= [1.37-2.63], p<0.001). Using the Programme de Medicalisation des Systemes Information (PMSI), a French cohort study reported the results of in-hospital mortality after colorectal resection, in France between 2009 and 2012. Of the 176,444 patients included, 35,586 had undergone SD surgery. The reported mortality after elective surgery for SD was 0.7%. Currently, mortality after prophylactic surgery for SD is less than 1%, ranging from 0.4% to 0.7%. From the American registry that included 2729 patients with SD operated on in emergency between 2012 and 2016, the latest published study reported an excess mortality of the Hartmann procedure compared with protected resection-anastomosis (7.6% vs. 2.9%, p= 0.011). However, as in all uncontrolled comparative studies, patients with Hartmann intervention were significantly more severe.

Morbidity after prophylactic colectomy has been reported in a large number of studies, but their exhaustive analysis is of limited interest due to the evolution of perioperative management (development of rehabilitation), the development of laparoscopic surgery and the time frame for analysis, which varies from study to study (30 or 90 days). Indeed, the type of complication reported varies considerably from one publication to another. For example, two monocentric series involving 500 and 576 patients respectively, who underwent laparoscopic SD surgery, reported a mortality rate of 0.2% and major complications in 11% of cases. The prevalence of anastomotic fistula was less than 2%. These figures for major morbidity of 10% were also found in a recent series in the literature (21,22). To figures from national databases, after adjustment for age, gender, ethnic origin, period of admission, and Charlson comorbidity score, compared with colon cancer, colectomy for SD was associated with an excess risk of post-operative infection (AOR, 1.67; 95% CI, 1.48-1.89; P .001) and stoma (AOR, 1.87; 95% CI, 1.65-2.11; P .001). In this study, the overall postoperative complication rate was impossible to determine, as each complication was detailed separately; on the other hand, the prevalence of stoma was high, being made in 7.55% of patients operated on for cold SD. Four years earlier, an analysis of the same database but focusing on patients operated on in 2001 and 2002 had been published, to compare the complication rates observed after an emergency or elective procedure. Emergency surgery was associated with higher morbidity and stoma rates (29% and 48.9%, respectively) than prophylactic colectomy (14.9% and 5.7%, respectively). It would appear interesting to know the rate of patients who will require a stoma during or after prophylactic colectomy for SD. Indeed, one of the major arguments in favor of prophylactic surgery is the risk of having to undergo emergency surgery in the event of a recurrence, with the provision of a stoma. In short, almost one patient in 6 (16%) will develop a complication after prophylactic colectomy for SD; the risk of the stoma may be as high as 6%. Few data are available on the prevalence of postoperative recurrence.

Clinical determinants linked to the patient, the causative pathology, and the surgical modalities have been identified in France as independent risk factors for postoperative mortality and morbidity. In contrast, few data are available in our healthcare system on the influence of non-clinical determinants such as socio-economic deprivation and territorial isolation. Several series suggest that socio-economic and territorial inequalities have an impact on postoperative morbidity and mortality for a large number of pathologies, such as cardiovascular disease, cancer, and obesity. Thus, patients from the most disadvantaged backgrounds are significantly more at risk of postoperative mortality and morbidity, particularly in the United States. However, socio-economic deprivation is a multidimensional concept that is difficult to grasp and measure. Several socio-economic indices have been developed, using medico-administrative data to which several indicators are applied (nationality, education, single-parent family, unemployment, access to housing, etc.).

In terms of postoperative morbidity, few data are available on the relationship between socio-economic deprivation and postoperative complications in colorectal surgery. While socio-economic deprivation significantly increased postoperative complications after ileostomy closure, this study included less than 100 patients. After left colectomy for cancer or diverticulitis, the prevalence of postoperative complications was significantly more frequent in the most disadvantaged patients (50.8 versus 41.2%, 0.0001) but only in univariate analysis. In the study of the Dutch registry, the absence of socio-economic deprivation represented an independent protective risk factor (risk relative to 0.7) of post-operative septic complications (i.e., anastomotic fistula abscess) after resection of colon cancer. To our knowledge, a single multicenter French study from the COINCIDE register evaluated the impact of socio-economic and territorial deprivation on morbidity and mortality in carcinological colorectal surgery, from a prospective multicentre COINCIDE database, which included other morbidity-related factors. From 2008 to 2010, 1259 curative colorectal resections were performed at AP-HP. In summary, after curative surgery for colorectal cancer, the most disadvantaged patients are 1.5 times more likely to develop severe postoperative complications. This risk is all the higher since they are men, aged 66 and over and operated by laparotomy of a rectal cancer. This study suggests that the determinants of health are multidimensional and are not limited to the performance of the healthcare system alone. The inclusion of this index in our surgical databases is therefore necessary, as is its use in health policy for resource allocation. To our knowledge, no study in the literature has assessed the impact of non-clinical determinants on the surgical management of SD. This French multicenter study aims to measure the impact of socio-economic and territorial inequalities on different aspects of surgical management by successively determining the prevalence of emergency surgery, access to minimally invasive surgery, postoperative morbidity and mortality, definitive stoma rate, and postoperative recurrence.

ELIGIBILITY:
Inclusion Criteria:

* - Patients aged over 18, operated on between 2010 and 2019, for sigmoid diverticulitis
* Patients aged 18 and over
* Patients undergoing emergency or elective surgery for sigmoid diverticulitis The patient was operated on between January 1, 2010, and December 31, 2019, with a follow-up of at least 3 months to determine morbi-mortality on the 90th postoperative day.

Exclusion Criteria:

* - Minor patient
* Surgical finding of colorectal cancer The patient operated on for diverticulitis of the right colon
* Patients with a history of chronic inflammatory bowel disease (Crohn's disease, hemorrhagic rectocolitis) and/or hereditary diseases predisposing to colorectal cancer (Lynch syndrome, familial polyposis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients aged over 18, operated on between 2010 and 2019, for sigmoid diverticulitis
  * Patients aged 18 and over
  * Patients undergoing emergency or elective surgery for sigmoid diverticulitis The patient was operated on between January 1, 2010, and December 31, 2019, with a follow-up of at least 3 months to determine morbi-mortality on the 90th postoperative day.
Sampling Method: Non-Probability Sample
Enrollment: 6800 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
90-day morbidity | From enrollment to the end of treatment at 90 days
90-day mortality | From enrollment to the end of treatment at 90 days

SECONDARY OUTCOMES:
- Prevalence of emergency versus prophylactic surgery and type of surgical procedure. | "From enrollment to the end of treatment at 90 days
  To assess the correlation between :
  * Prevalence of emergency versus prophylactic surgery and type of surgical procedure.
  * Index of socio-economical deprivation (EDI)
Prevalence of minimally invasive surgery (laparoscopy, robot) versus laparotomy surgery | "From enrollment to the end of treatment at 90 days
  To assess the correlation between :
  Prevalence of minimally invasive surgery (laparoscopy, robot) versus laparotomy surgery
  - Index of socio-economical deprivation
- Prevalence of definitive stoma | "From enrollment to the end of treatment at 90 days
  To assess the correlation between :
  * - Prevalence of definitive stoma
  * Index of socio-economical deprivation (EDI)
Prevalence of postoperative recurrence | "From enrollment to the end of treatment at 90 days
  To assess the correlation between :
  * Prevalence of postoperative recurrence
  * Index of socio-economical deprivation (EDI)

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No